CLINICAL TRIAL: NCT04178772
Title: Characterizing Successful Myopic Multifocal Contact Lens Wearers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: To ensure the safety of participants during the COVID-19 pandemic, this clinical trial is suspended until further notice. This study was terminated due to the lockdown requirements.
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-5945
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Results first posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- JJVC Marketed Contact Lens (Experimental): Eligible subjects that have no experience with soft multifocal lenses for more than 2 years will be assigned to a single study lens type worn in both eyes daily for at least 6 hours per day, everyday for approximately 12 weeks.
  Interventions: Device: Acuvue Moist Multifocal Contact Lens JJVC Marketed Contact Lens

INTERVENTIONS:
Device: Acuvue Moist Multifocal Contact Lens JJVC Marketed Contact Lens — JJVC Marketed Contact Lens

SUMMARY:
This will be a prospective, single group, single-arm, and bilateral dispensing study. Subjects will be assigned to a single study lens type to be worn bilaterally in daily wear, and daily disposable modality, for at least 6 hours per day every day for approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Potential Subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The participant must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Is at least 40 years of age (inclusive) at the time of screening and has full legal capacity to volunteer.
  4. Had a self-reported eye examination in the last two years.
  5. The subject must either already be wearing a presbyopic correction (e.g., reading spectacles over contact lenses, or multifocal spectacles, etc.) or respond positively to at least one symptom on the 'Presbyopic Symptoms Questionnaire".
  6. Can achieve best corrected distance monocular visual acuity of at least +0.20 logMAR and binocular visual acuity of at least +0.10 logMAR with refraction.
  7. Have a refractive cylinder of ≤1.00 D in each eye.
  8. Has corrected best sphere equivalent distance refraction in the range -0.50 D of -6.00 D in each eye (vertex corrected if greater than -4.00D).
  9. Have a reading ADD power in the range of +0.75 D to +1.75 D (inclusive) in each eye.
  10. Have a wearable pair of spectacles (at the discretion of the investigator) to wear when they cannot wear the study lenses.

      Exclusion Criteria:
* Potential Subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Participation in any contact lens or lens care clinical trial within 1 week prior to study enrollment.
  2. Employee or immediate family member of an employee of the Centre for Ocular Research & Education listed on the study Delegation Log (e.g., Investigator, Coordinator, Technician).
  3. Is currently pregnant or lactating, by self-report, or planning a pregnancy at the time of enrollment.
  4. Has any known active ocular disease and/or allergies, ocular infections or other abnormalities that are known to interfere with contact lens wear (at the discretion of the investigator). This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or corneal distortion.
  5. Is using any topical ocular medications other than lubricating eye drops.
  6. Known to have any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease.
  7. Have any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear (at the discretion of the investigator). This may include, but not be limited to, hyperthyroidism, recurrent herpes simplex/zoster, Sjogren's syndromes, xerophthalmia, acne rosacea, Stevens-Johnson syndromes.
  8. Had a diagnosis of a condition known to affect ocular prescription or ocular surface or tear film e.g., rheumatoid arthritis, diabetes.
  9. Had a change within the previous 3 months to the dosage of a systemic medication known to affect ocular prescription or ocular surface or tear film (e.g., steroids) that in the opinion of the investigator may affect a study outcome variable.
  10. Has undergone cataract or refractive error surgery (e.g., radial keratotomy, PRK, LASIK, etc.), or has any planned (during the study) major surgery (e.g. hip replacement), or any planned ocular surgery (e.g. cataract or refractive error surgery).
  11. Is a current rigid contact lens wearer, or is wearing contact lenses on extended wear basis, or has a history of extended wear in the past 6 months.
  12. Has worn soft MF CLs in the past 2 years or is a habitual wearer of monovision CLs.
  13. Has a constant unilateral strabismus at both far and near distances, or has anisometropia >2 D between both eyes, or has amblyopia.
  14. Has a known sensitivity to the diagnostic pharmaceuticals to be used in the study (Refresh Plus® rewetting drop solution, Sodium Fluorescein or Alcon Clear Care Cleaning System).
  15. Has any Grade 3.0 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the biomicroscopy classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear (at the discretion of the investigator).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- Centre for Ocular Research and Education, University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 29 subjects were enrolled into this study. Of those enrolled, 27 were dispensed study lenses, while 2 subjects failed to meet all eligibility criteria. Of those dispensed, 19 completed the study while 8 subjects were discontinued. This study was terminated early due to COVID-19.
Groups:
- Etafilcon A Multifocal Lens: Subjects that wore the etafilcon A lens during any point of the study.
Period: Overall Study
Arm/Group | Etafilcon A Multifocal Lens
Started | 27
Completed | 19
Not Completed | 8
Not completed — Unsatisfacotry VIsual Response | 1
Not completed — study terminated early due to COVID-19 | 7

BASELINE CHARACTERISTICS:
Population: All subjects dispensed in a study lens.
Groups:
- Dispensed Subject: All subjects dispensed a study lens.
Arm/Group | Dispensed Subject
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (3.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 2
  White | 24
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 27

OUTCOME MEASURES:

1. Primary Outcome: Quest Questionnaire Classification Summary
Description: Subjects are classified into 1 of 4 mutually exclusive groups based on their responses to 6 individual items. 5 items were assessed using the 7-point like-rt scale. A composite score "Life Satisfaction" was calculated for each subject by summing their responses, the final score ranges 0-35 points. Where higher scores indicate higher satisfaction with life. The final item was assessed using a 5 point like-rt scale. If a subject scored 26 or higher for the composite score and responded positively (4 or 5) to the final item, then a subject was classified as "Content & Driven". If a subject scored 26 or higher but did not respond positively, then "Content & Indifferent". If a subject scored lower than 26 and responded positively, then "Discontented & Driven". Lastly, if a subject scored lower than 26 but did not respond positively, then "Discontented & Indifferent". The percentage of subjects for each group was reported.
Time Frame: Baseline
Population: All subjects dispensed a study lens.
Measure: Number; unit: Percentage of Participants
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
Percentage of Participants
  Discontented & Driven | 22.2
  Content & Driven | 33.3
  Discontented & Indifferent | 11.2
  Content & Indifferent | 33.3

2. Primary Outcome: Proportion of Successful Lens Wearers
Description: Successful lens wearers were defined as subjects that fit the following criteria: 1.Completed all required study visits, 2. responded Excellent or Very Good to both the individual questionnaire items (Overall quality of vision and Overall Comfort) and 3. the investigator would recommend the study lenses. Overall quality of Vision and Overall Comfort are individual questionnaire items with the response set of 0: Not Applicable, 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor. Investigator recommendation was determined by the individual item "In your opinion, is it suitable to prescribe contact lenses for this subject? (Yes/No)". The proportion of successful lens wearers was reported.
Time Frame: 12-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Number; unit: Proportion of Participants
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
Proportion of Participants | 0.593

3. Secondary Outcome: Monocular Contrast Threshold
Description: Monocular Contrast threshold was measured at Distance (4 meter) for both the left and right eyes using the M&S clinical trial suit (CTS) under standard room illumination. Contrast threshold was collected at Baseline, post lens fitting, 2-week follow-up evaluation and the 12-week evaluation. Contrast threshold at baseline was measured while wearing a spherical-cylinder refraction in a trial frame. The M&S system displayed the contrast threshold score in log units. The average contrast threshold was reported for each timepoint.
Time Frame: Baseline, Post Lens Fitting, 2-Week Follow-up, 12-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: log CS
Units Other Than Participants: eyes
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
Number analyzed (eyes) | 54
log CS
  Baseline | -1.32 (0.174)
  Post Lens Fitting: number analyzed (Participants) | 24
  Post Lens Fitting: number analyzed (eyes) | 48
  Post Lens Fitting | -1.15 (0.244)
  2-Week Follow-up: number analyzed (Participants) | 23
  2-Week Follow-up: number analyzed (eyes) | 46
  2-Week Follow-up | -1.24 (0.196)
  12-Week Follow-up: number analyzed (Participants) | 9
  12-Week Follow-up: number analyzed (eyes) | 18
  12-Week Follow-up | -1.16 (0.226)

4. Secondary Outcome: Binocular Contrast Threshold
Description: Binocular Contrast threshold was measured at Distance (4 meter) using the M&S clinical trial suit (CTS) under standard room illumination. Contrast threshold was collected at Baseline, post lens fitting, 2-week follow-up evaluation and the 12-week evaluation. Contrast threshold at baseline was measured while wearing a spherical-cylinder refraction in a trial frame. The M&S system displayed the contrast threshold score in log units.
Time Frame: Baseline, Post Lens Fitting, 2-Week Follow-up, 12-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: log CS
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
log CS
  Baseline | -1.46 (0.178)
  Post Lens Fitting: number analyzed (Participants) | 24
  Post Lens Fitting | -1.32 (0.228)
  2-Week Follow-up: number analyzed (Participants) | 23
  2-Week Follow-up | -1.43 (0.196)
  12-Week Follow-up: number analyzed (Participants) | 9
  12-Week Follow-up | -1.35 (0.209)

5. Secondary Outcome: Photopic Pupillometry
Description: Pupillometry was measured for both the left and right eyes at baseline and the 1-week follow-up evaluation . Pupil size was measured at distance, intermediate and near positions under photopic (500 lux) conditions using the NeurOptic VIP-300 pupilometer. The average pupil size across both eyes was reported for each distance and timepoint.
Time Frame: Baseline, 1-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
mm
  Baseline: Distance (4 meter) | 3.85 (0.578)
  Baseline: Intermediate (1 meter) | 3.73 (0.568)
  Baseline: Near (40 cm) | 3.70 (0.608)
  1-Week Follow-up: Distance (4 meter): number analyzed (Participants) | 24
  1-Week Follow-up: Distance (4 meter) | 3.87 (0.502)
  1-Week Follow-up: Intermediate (1 meter): number analyzed (Participants) | 24
  1-Week Follow-up: Intermediate (1 meter) | 3.64 (0.428)
  1-Week Follow-up: Near (40 cm): number analyzed (Participants) | 24
  1-Week Follow-up: Near (40 cm) | 3.44 (0.463)

6. Secondary Outcome: Scotopic Pupillometry
Description: Pupillometry was measured for both the left and right eyes at baseline and the 1-week follow-up evaluation . Pupil size was measured at distance, intermediate and near positions under scotopic (0 lux) conditions using the NeurOptic VIP-300 pupilometer. The average pupil size across both eyes was reported for each distance and timepoint.
Time Frame: Baseline, 1-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
mm
  Baseline: Distance (4 meter) | 5.92 (0.804)
  Baseline: Intermediate (1 meter) | 5.75 (0.786)
  Baseline: Near (40 cm) | 5.33 (0.816)
  1-Week Follow-up: Distance (4 meter): number analyzed (Participants) | 24
  1-Week Follow-up: Distance (4 meter) | 5.79 (0.872)
  1-Week Follow-up: Intermediate (1 meter): number analyzed (Participants) | 24
  1-Week Follow-up: Intermediate (1 meter) | 5.65 (0.769)
  1-Week Follow-up: Near (40 cm): number analyzed (Participants) | 24
  1-Week Follow-up: Near (40 cm) | 5.19 (0.839)

7. Secondary Outcome: Near Stereopsis Threshold
Description: Near Stereopsis threshold was collected binocularly using a Randot Stereopsis book at near (40cm) at baseline (over bare eyes), and at 10-minutes post lens fitting, 2-Week and 12-week follow-up evaluations over the study contact lenses. The average stereopsis threshold for each timepoint was reported.
Time Frame: Baseline, 10-mintue Post Lens Fitting, 2-Week Follow-up, 12-Week Follow-up
Population: All subjects enrolled the study.
Measure: Mean (Standard Deviation); unit: seconds of arc
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 28
seconds of arc
  Baseline | 43.04 (17.968)
  10-minutes Post Lens Fitting: number analyzed (Participants) | 24
  10-minutes Post Lens Fitting | 58.54 (51.213)
  2-Week Follow-up: number analyzed (Participants) | 23
  2-Week Follow-up | 43.48 (16.544)
  12-Week Follow-up: number analyzed (Participants) | 9
  12-Week Follow-up | 41.67 (14.577)

8. Secondary Outcome: Blur Tolerance
Description: Blur tolerance was assessed by subjects being presented with a series on images on a screen. Two aspects of blur were evaluated, noticeable blur and objectionable blur; where, noticeable blur was defined as the threshold in diopters at which point the subject indicated a "just noticeable blur", while objectional blur was defined as the point which the subject indicated the blur of the image to be "absolutely intolerable". Blur tolerance was measured binocularly at 1-meter at baseline only.
Time Frame: Baseline
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
diopters
  Noticeable blur | 0.2 (0.06)
  Objectionable blur | 0.3 (0.07)

9. Secondary Outcome: Fixation Disparity With Refraction
Description: Fixation disparity with Refraction was measured at baseline with a Mallet Unit for both distance (4 meter) and near (40 cm). This test measures small misalignments between eyes when the eyes are in a fused state. The average amount of base (prism diopters) was reported. The Amount of base can range from 0.00 to 4.00.
Time Frame: Baseline
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
prism diopters
  Distance | 0.74 (1.130)
  Near | 0.63 (1.079)

10. Secondary Outcome: Non-invasive Tear Break-up Time
Description: Measurement of non-invasive tear break up time (NITBUT) was conducted using a Placido disc topographer in both the left and right eyes on a bare eye at baseline and over the study contact lens 10 minutes post-lens insertion and at the 2-Week follow-up evaluation. Subjects were instructed to blink three times and then hold their eyes open. At the hold time was started, time was stopped once the first area of distortion or break in the tear film was observed. Three replicates were taken on each eye. The average NITBUT across eyes and replicate at each time point was provided. Larger values of NITBUT indicates better tear film.
Time Frame: Baseline, 10-minute Post Lens Fitting, 2-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
Number analyzed (eyes) | 54
seconds
  Baseline | 5.99 (3.839)
  10 minutes Post-Lens Insertion: number analyzed (Participants) | 24
  10 minutes Post-Lens Insertion: number analyzed (eyes) | 48
  10 minutes Post-Lens Insertion | 3.75 (1.241)
  2-Week Follow-up: number analyzed (Participants) | 23
  2-Week Follow-up: number analyzed (eyes) | 46
  2-Week Follow-up | 3.88 (1.667)

11. Secondary Outcome: Coma
Description: Coma was measured over 2 seconds after blink in both the left and right eyes at baseline (over bare eye) and at 10-minutes post-lens fitting, 2-week, and 12-week follow-up evaluations over the study contact lenses using the COAS wavefront sensor. Both vertical and horizontal Coma was collected in each eye. The average vertical and horizontal coma at each timepoint was reported.
Time Frame: Baseline, 10-minute Post Lens Fitting, 2-Week Follow-up, 12-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: eyes
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
Number analyzed (eyes) | 54
microns
  Horizontal: Baseline | 0.02 (0.045)
  Horizontal: 10 minutes Post-Lens Insertion: number analyzed (Participants) | 24
  Horizontal: 10 minutes Post-Lens Insertion: number analyzed (eyes) | 48
  Horizontal: 10 minutes Post-Lens Insertion | 0.03 (0.062)
  Horizontal: 2-Week Follow-up: number analyzed (Participants) | 23
  Horizontal: 2-Week Follow-up: number analyzed (eyes) | 46
  Horizontal: 2-Week Follow-up | 0.03 (0.066)
  Horizontal: 12-Week Follow-up: number analyzed (Participants) | 9
  Horizontal: 12-Week Follow-up: number analyzed (eyes) | 18
  Horizontal: 12-Week Follow-up | 0.03 (0.076)
  Vertical: Baseline | 0.02 (0.047)
  Vertical: 10 minutes Post-Lens Insertion: number analyzed (Participants) | 24
  Vertical: 10 minutes Post-Lens Insertion: number analyzed (eyes) | 48
  Vertical: 10 minutes Post-Lens Insertion | 0.03 (0.054)
  Vertical: 2-Week Follow-up: number analyzed (Participants) | 23
  Vertical: 2-Week Follow-up: number analyzed (eyes) | 46
  Vertical: 2-Week Follow-up | 0.02 (0.054)
  Vertical: 12-Week Follow-up: number analyzed (Participants) | 9
  Vertical: 12-Week Follow-up: number analyzed (eyes) | 18
  Vertical: 12-Week Follow-up | 0.01 (0.080)

12. Secondary Outcome: Higher Order Aberration
Description: Higher Order Aberration (HOA) was measured over 2 seconds after blink in both the left and right eyes at baseline (over bare eye) and at 10-minutes post-lens fitting, 2-week, and 12-week follow-up evaluations over the study contact lenses using the COAS wavefront sensor. The average HOA at each timepoint was reported.
Time Frame: Baseline, 10-minute Post Lens Fitting, 2-Week Follow-up, 12-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: eyes
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
Number analyzed (eyes) | 54
microns
  Baseline | 0.17 (0.044)
  10 minutes Post-Lens Insertion: number analyzed (Participants) | 24
  10 minutes Post-Lens Insertion: number analyzed (eyes) | 48
  10 minutes Post-Lens Insertion | 0.21 (0.146)
  2-Week Follow-up: number analyzed (Participants) | 23
  2-Week Follow-up: number analyzed (eyes) | 46
  2-Week Follow-up | 0.23 (0.207)
  12-Week Follow-up: number analyzed (Participants) | 9
  12-Week Follow-up: number analyzed (eyes) | 18
  12-Week Follow-up | 0.21 (0.060)

13. Secondary Outcome: Keratometry (Diopters)
Description: Keratometry (corneal curvature) collected at baseline for each eye (left and right) using an autokeratometer. The measurement was recorded in diopters (DK) of major keratometric meridians. The average of each measurement was reported.
Time Frame: Baseline
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: eyes
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
Number analyzed (eyes) | 54
diopters
  Steep | 44.46 (1.628)
  Flat | 43.72 (1.735)

14. Secondary Outcome: Keratometry (Degrees)
Description: Keratometry (corneal curvature) collected at baseline for each eye (left and right) using an autokeratometer. The measurement was recorded for locations (degrees) of major keratometric meridians. The average of each measurement was reported.
Time Frame: Baseline
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: eyes
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
Number analyzed (eyes) | 54
degrees
  Steep | 86.43 (21.576)
  Flat | 106.43 (74.425)

15. Secondary Outcome: Objective Accommodation With Distance Refraction
Description: Objective accommodation with sphero-cylindrical distance refraction was collected using the WAM-5500 auto-refractor at distance (4-meter), Intermediate (1-meter) and Near (40cm) in both the left and right eyes at baseline, 10-minutes post lens fitting, 2-week and 12-week follow-up evaluations. Measurements at baseline were collected on bare eyes and over the study contact lens at the follow-up evaluations. The average sphere power (diopters) across eyes was report for each distance and timepoint.
Time Frame: Baseline, 10-minute Post Lens Fitting, 2-Week Follow-up, 12-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: eyes
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
Number analyzed (eyes) | 54
diopters
  Distance: Baseline | 0.61 (0.400)
  Distance: 10-Minutes Post Lens Fitting: number analyzed (Participants) | 24
  Distance: 10-Minutes Post Lens Fitting: number analyzed (eyes) | 48
  Distance: 10-Minutes Post Lens Fitting | 0.17 (0.347)
  Distance: 2-Week Follow-up: number analyzed (Participants) | 23
  Distance: 2-Week Follow-up: number analyzed (eyes) | 46
  Distance: 2-Week Follow-up | 0.15 (0.296)
  Distance: 12-Week Follow-up: number analyzed (Participants) | 9
  Distance: 12-Week Follow-up: number analyzed (eyes) | 18
  Distance: 12-Week Follow-up | 0.11 (0.296)
  Intermediate: Baseline | 0.35 (0.450)
  Intermediate: 10-Minutes Post Lens Fitting: number analyzed (Participants) | 24
  Intermediate: 10-Minutes Post Lens Fitting: number analyzed (eyes) | 48
  Intermediate: 10-Minutes Post Lens Fitting | -0.09 (0.343)
  Intermediate: 2-Week Follow-up: number analyzed (Participants) | 23
  Intermediate: 2-Week Follow-up: number analyzed (eyes) | 46
  Intermediate: 2-Week Follow-up | -0.06 (0.366)
  Intermediate: 12-Week Follow-up: number analyzed (Participants) | 9
  Intermediate: 12-Week Follow-up: number analyzed (eyes) | 18
  Intermediate: 12-Week Follow-up | -0.11 (0.335)
  Near: Baseline | -0.24 (0.684)
  Near: 10-Minutes Post Lens Fitting: number analyzed (Participants) | 24
  Near: 10-Minutes Post Lens Fitting: number analyzed (eyes) | 48
  Near: 10-Minutes Post Lens Fitting | -0.57 (0.509)
  Near: 2-Week Follow-up: number analyzed (Participants) | 23
  Near: 2-Week Follow-up: number analyzed (eyes) | 46
  Near: 2-Week Follow-up | -0.60 (0.596)
  Near: 12-Week Follow-up: number analyzed (Participants) | 9
  Near: 12-Week Follow-up: number analyzed (eyes) | 18
  Near: 12-Week Follow-up | -0.61 (0.407)

16. Secondary Outcome: Binocular Visual Acuity (logMAR)
Description: Binocular Visual Acuity (logMAR) was collected using logMAR visual acuity chart under standard room illumination at distance (4 meter), intermediate (64cm) and near (40cm) at 10 minutes-post lens fitting, and the 1-, 2-, 6- and 12-week follow-up evaluations. However, intermediate was not collected post fitting and at the 1-week follow-up evaluation. A value of 0.0 logMAR is approximate to 20/20 Snellen Visual Acuity. Lower values of visual acuity (logMAR) indicate better vision. The average visual acuity was reported for each distance and timepoint.
Time Frame: 10-minute Post Lens Fitting, 1-Week Follow-up, 2-Week Follow-up, 6-Week Follow-up, 12-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
logMAR
  Distance: 10-Minutes Post Lens Fitting | -0.076 (0.0719)
  Distance: 1-Week Follow-up: number analyzed (Participants) | 24
  Distance: 1-Week Follow-up | -0.104 (0.0646)
  Distance: 2-Week Follow-up: number analyzed (Participants) | 23
  Distance: 2-Week Follow-up | -0.102 (0.0741)
  Distance: 6-Week Follow-up: number analyzed (Participants) | 19
  Distance: 6-Week Follow-up | -0.107 (0.0681)
  Distance: 12-Week Follow-up: number analyzed (Participants) | 9
  Distance: 12-Week Follow-up | -0.098 (0.0570)
  Near: 10-Minutes Post Lens Fitting | -0.012 (0.1013)
  Near: 1-Week Follow-up: number analyzed (Participants) | 24
  Near: 1-Week Follow-up | -0.024 (0.1091)
  Near: 2-Week Follow-up: number analyzed (Participants) | 23
  Near: 2-Week Follow-up | -0.051 (0.1019)
  Near: 6-Week Follow-up: number analyzed (Participants) | 19
  Near: 6-Week Follow-up | -0.077 (0.0922)
  Near: 12-Week Follow-up: number analyzed (Participants) | 9
  Near: 12-Week Follow-up | -0.027 (0.1196)
  Intermediate: 2-Week Follow-up: number analyzed (Participants) | 23
  Intermediate: 2-Week Follow-up | -0.152 (0.0725)
  Intermediate: 6-Week Follow-up: number analyzed (Participants) | 19
  Intermediate: 6-Week Follow-up | -0.166 (0.0476)
  Intermediate: 12-Week Follow-up: number analyzed (Participants) | 9
  Intermediate: 12-Week Follow-up | -0.131 (0.0549)

17. Secondary Outcome: Monocular Visual Acuity (logMAR)
Description: Monocular Visual Acuity (logMAR) was collected in both the left and right eyes using logMAR visual acuity chart under standard room illumination at distance (4 meter), intermediate (64cm) and near (40cm) at 10 minutes-post lens fitting, and the 1-, 2-, 6- and 12-week follow-up evaluations. However, intermediate was not collected post fitting and at the 1-week follow-up evaluation. A value of 0.0 logMAR is approximate to 20/20 Snellen Visual Acuity. Lower values of visual acuity (logMAR) indicate better vision. The average visual acuity was reported for each distance and timepoint.
Time Frame: 10-minute Post Lens Fitting, 1-Week Follow-up, 2-Week Follow-up, 6-Week Follow-up, 12-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Etafilcon A Multifocal Lens
Number analyzed (Participants) | 27
Number analyzed (eyes) | 54
logMAR
  Distance: 10-Minutes Post Lens Fitting | -0.013 (0.0828)
  Distance: 1-Week Follow-up: number analyzed (Participants) | 24
  Distance: 1-Week Follow-up: number analyzed (eyes) | 48
  Distance: 1-Week Follow-up | -0.034 (0.0808)
  Distance: 2-Week Follow-up: number analyzed (Participants) | 23
  Distance: 2-Week Follow-up: number analyzed (eyes) | 46
  Distance: 2-Week Follow-up | -0.038 (0.0774)
  Distance: 6-Week Follow-up: number analyzed (Participants) | 19
  Distance: 6-Week Follow-up: number analyzed (eyes) | 38
  Distance: 6-Week Follow-up | -0.040 (0.0790)
  Distance: 12-Week Follow-up: number analyzed (Participants) | 9
  Distance: 12-Week Follow-up: number analyzed (eyes) | 18
  Distance: 12-Week Follow-up | -0.024 (0.0708)
  Near: 10-Minutes Post Lens Fitting | 0.082 (0.1060)
  Near: 1-Week Follow-up: number analyzed (Participants) | 24
  Near: 1-Week Follow-up: number analyzed (eyes) | 48
  Near: 1-Week Follow-up | 0.063 (0.1185)
  Near: 2-Week Follow-up: number analyzed (Participants) | 23
  Near: 2-Week Follow-up: number analyzed (eyes) | 46
  Near: 2-Week Follow-up | 0.019 (0.0975)
  Near: 6-Week Follow-up: number analyzed (Participants) | 19
  Near: 6-Week Follow-up: number analyzed (eyes) | 38
  Near: 6-Week Follow-up | 0.021 (0.0899)
  Near: 12-Week Follow-up: number analyzed (Participants) | 9
  Near: 12-Week Follow-up: number analyzed (eyes) | 18
  Near: 12-Week Follow-up | 0.029 (0.1039)
  Intermediate: 2-Week Follow-up: number analyzed (Participants) | 23
  Intermediate: 2-Week Follow-up: number analyzed (eyes) | 46
  Intermediate: 2-Week Follow-up | -0.074 (0.0826)
  Intermediate: 6-Week Follow-up: number analyzed (Participants) | 19
  Intermediate: 6-Week Follow-up: number analyzed (eyes) | 38
  Intermediate: 6-Week Follow-up | -0.095 (0.0657)
  Intermediate: 12-Week Follow-up: number analyzed (Participants) | 9
  Intermediate: 12-Week Follow-up: number analyzed (eyes) | 18
  Intermediate: 12-Week Follow-up | -0.064 (0.0721)

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 3 months per subject.
Arm/Group | Etafilcon A Multifocal Lens
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT04178772/Prot_SAP_000.pdf